CLINICAL TRIAL: NCT03585517
Title: Safety and Efficacy Evaluation of IM23 CAR-T Cells On CD123+ AML Patients
Brief Title: Safety and Efficacy Evaluation of IM23 CAR-T Cells (IM23CAR-T)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Immunochina Medical Science & Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YMCART201806
Record Dates: First submitted 2018-07-01; First posted 2018-07-13 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2018-07

CONDITIONS: AML

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IM23 CART (Experimental): All patients will be treated with fludarabine and cyclophosphamide for 3 days,then,CAR-T cells expressing CD123 CAR will be infused 24-96 hours later.
  Interventions: Drug: IM23

INTERVENTIONS:
Drug: IM23 — T Cells Expressing an Anti-CD123 Chimeric Antigen Receptor

SUMMARY:
Assessment of the Safety and Feasibility of Administering T Cells Expressing an Anti-CD123 Chimeric Antigen Receptor to Patients With CD123+ AML

DETAILED DESCRIPTION:
Assessment of the Safety and Feasibility of Administering T Cells Expressing an Anti-CD123 Chimeric Antigen Receptor to Patients With CD123+ AML and determine the best dosage.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CD123+ Refractory or Relapsed AML
* To be aged 3 to 80 years
* Expression of CD123 in Blast ≥90%
* ECOG score ≤2
* Voluntary participation in the clinical trials and sign the informed consent.

Exclusion Criteria:

* Intracranial hypertension or unconsciousness
* Respiratory failure
* CD19 negative
* Disseminated intravascular coagulation
* ALT /AST>3 x normal value; Creatinine> 1.5 x normal value; Bilirubin >2.0 x -normal value
* Hematosepsis or Uncontrolled active infection
* Uncontrolled diabetes
* Abalienation;
* Patients in pregnancy or breast-feeding period
* Previously treatment with any gene therapy products
* Any uncontrolled medical disorders that the researchers consider are not eligible to participate the clinical trial

Ages: 3 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-07-21 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of study related adverse events | 2 years
  defined as >= Grade 3 signs/symptoms, laboratory toxicities, and clinical events) that are possibly, likely, or definitely related to study treatment Adverse events assessed according to NCI-CTCAE v4.0 criteria 2

CONTACTS AND LOCATIONS:
Locations (1):
- Xian Lu, Beijing, China